CLINICAL TRIAL: NCT03632837
Title: HaemoAdsorption Nach Reanimation An ECMO
Acronym: HANRAE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: CytoSorbents Corporation and CytoSorbents Medical Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UKEHANRAE
Record Dates: First submitted 2018-05-03; First posted 2018-08-16 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Cardiac Arrest; Resuscitation; Inflammation; Multi-Organ Disorder
Keywords: extracorporal circulation; hemoadsorption; post resuscitation syndrome
MeSH Terms: conditions — Heart Arrest; Inflammation

STUDY DESIGN:
Masking Description: Participants are regularily going to be unconsciuos during the differential treatment phase due to the nature and severity of their condition, yet exceptions to this are not going to be suppressed for obvious ethical reasons.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Treatment (Experimental): Inclusion of an extracorporal in line adsorbing cartridge for 48h (with a cartridge exchange at 24h) post establishing ECMO in addition to standard post resuscitation intensive care
  Interventions: Device: Hemoadsorption
- Control (No Intervention): ECMO and standard post resuscitation intensive care without any additional module in extracorporal circulation

INTERVENTIONS:
Device: Hemoadsorption — see arm description
  Arms: Treatment

SUMMARY:
This study evaluates the use of an additional hemoadsorption device in adult patients undergoing veno-arterial extracorporal membrane oxygenation (ECMO) following cardiac arrest and cardiopulmonary resuscitation in respect to its effects on post resuscitation inflammatory syndrome.

At implantation of the ECMO the participants are going to be randomized into a treatment and a control group. The first will be outfitted with a polymer-based adsorption device implemented in the extracorporal circulation established by ECMO for 48h, the control group is going to be treated by ECMO and standard intensive care alone. To detect any significant differences in terms of inflammatory response and patient outcome the investigators will regularly determine the blood levels of certain cytokines in fixed intervalls. In addition, the investigators are going to compare secondary clinical outcome parameters like organ disfunction and 30d mortality.

DETAILED DESCRIPTION:
Even after successful return of spontaneus circulation (ROSC), patients suffering a cardiac arrest with subsequent cardipulmonary resuscitation (CPR) are still facing a significant morbidity and mortality in the post-resuscitation phase. They are nowadays often subjected to extracorporal membrane oxygenation (ECMO), supplementing or even replacing cardiac and/or pulmonary function for a certain period in order to reduce the workload for these critical organs. However, as well as the initial ischemia/reperfusion damage, subsequent procedures create significant stress to the patients organism, causing severe inflammation and contributing to post-resuscitation single or multiple organ disfunction and/or failure.

Continously eliminating relevant mediators of inflammation by adsorption to a polymer-based material in extracorporal circulation has been shown to influence the course of this inflammatory syndrome in patients with severe infection and sepsis. Any relevant clinical studies evaluating the use of such a device in post-resuscitation care are still lacking, yet.

Therefore, in this study the investigators are going to test the hypothesis that such a device is capable of significantly altering the cytokine levels during and even shortly after a 48h treatment period in addition to the standard ECMO therapy all patients are going to receive. As a secondary outlook, the investigators are going to compare the clinical outcome of the patients in terms of major organ disfunction and overall 30d mortality.

At the time extracoporal circulation is established during or after CPR, all participants (n=40) are enrolled and randomized into a treatment and a control group. The extracorporal circulation over the ECMO device is then outfitted with a certified in line adsorption cartridge for the treatment group. Due to technical reasons, this cartridge has to be exchanged for another identical module after 24h of continuous treatment. Adsorption therapy is terminated after 48h. The control group is subjected to ECMO without any additional modules. Both groups are receiving standard intensive care during the course of the study. All diagnostic and therapeutic decisions with the exemption of those directly concerning the hemoadsorption and sampling protocol are at sole discretion of the clinical staff.

For both groups, blood samples are taken at time points 0,6,12,24,36,48,72h after establishment of ECMO or time of death, respectively. Relevant parameters are then determined in different diagnostic and research laboratories with/without sample preprocessing by the study personal in accordance with preanalytic requirements. All relevant clinical data is extracted from the digital patient data management system (PDMS).

ELIGIBILITY:
All patients receiving a veno-arterial ECMO after cardiac arrest at the study site are eligible for the study. Thus, the criteria are defined by the SOP "ECMO bei Reanimation" of the University Heart Center Hamburg:

Inclusion Criteria:

* observed cardiac arrest with initial hyperdynamic rhythm and sufficient primary resuscitation

Exclusion Criteria (absolute):

* existing "do-not-resuscitate"-order from the patient/a priori palliative situation
* severe trauma
* severe acute bleeding due to any cause
* confirmed or highly likely relevant and severe persistent neurologic impairment
* severe limiting comorbidities with independent and relevant reduction of life expectancy (e.g. malignoma, preexistent heart failure syndrome, obstructive/restrictive lung disease, hepatic cirrhosis)

Exclusion Criteria (relative, at the discretion of the responsible provider):

* severe initial lacacidosis
* prolongued mechanical resuscitation (>30min)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
IL-6 at hour 6 | 6 hours post establishment of extracorporal membrane oxygenation (ECMO)
  Blood levels of interleukine 6 will be compared between intervention and control group
IL-6 at hour 12 | 12 hours post establishment of extracorporal membrane oxygenation (ECMO)
  Blood levels of interleukine 6 will be compared between intervention and control group
IL-6 at hour 24 | 24 hours post establishment of extracorporal membrane oxygenation (ECMO)
  Blood levels of interleukine 6 will be compared between intervention and control group
IL-6 at hour 48 | 48 hours post establishment of extracorporal membrane oxygenation (ECMO)
  Blood levels of interleukine 6 will be compared between intervention and control group
IL-6 at hour 72 | 72 hours post establishment of extracorporal membrane oxygenation (ECMO)
  Blood levels of interleukine 6 will be compared between intervention and control group
TNF-a at hour 6 | 6 hours post establishment of extracorporal membrane oxygenation (ECMO)
  Blood levels of human tumor necrosis factor alpha will be compared between intervention and control group
TNF-a at hour 12 | 12 hours post establishment of extracorporal membrane oxygenation (ECMO)
  Blood levels of human tumor necrosis factor alpha will be compared between intervention and control group
TNF-a at hour 24 | 24 hours post establishment of extracorporal membrane oxygenation (ECMO)
  Blood levels of human tumor necrosis factor alpha will be compared between intervention and control group
TNF-a at hour 48 | 48 hours post establishment of extracorporal membrane oxygenation (ECMO)
  Blood levels of human tumor necrosis factor alpha will be compared between intervention and control group
TNF-a at hour 72 | 72 hours post establishment of extracorporal membrane oxygenation (ECMO)
  Blood levels of human tumor necrosis factor alpha will be compared between intervention and control group

SECONDARY OUTCOMES:
S1P | at hours 0,6,12,24,48,72 post establishment of extracorporal membrane oxygenation (ECMO)
  Blood levels of sphingosine-1-phosphate will be compared between intervention and control group.
PCT | at hours 0,6,12,24,48,72 post establishment of extracorporal membrane oxygenation (ECMO)
  The serum levels of procalcitonine will be compared between intervention and control group.
CRP | at hours 0,6,12,24,48,72 post establishment of extracorporal membrane oxygenation (ECMO)
  The plasma levels of C-related peptide will be compared between intervention and control group.
Leukocytes | at hours 0,6,12,24,48,72 post establishment of extracorporal membrane oxygenation (ECMO)
  The number of leukocytes in simple blood count will be compared between intervention and control group.
BNP | at hours 0,6,12,24,48,72 post establishment of extracorporal membrane oxygenation (ECMO)
  The serum levels of n-terminal pro brain natriuretic peptide will be compared between intervention and control group.
Mean arterial pressure (MAP) | Continuosly from enrollment to 72h post.
  The mean arterial pressure as calculated automatically from the invasively measured arterial pressure curve will be compared between intervention and control group.
Heart rate (HR) | Continuosly from enrollment to 72h post.
  The continuously monitored heart rate will be compared between intervention and control group.
Central venous pressure (CVP) | Continuosly from enrollment to 72h post.
  The continuously and invasively measured mean central venous pressure will be compared between intervention and control group, if available.
haemodynamically relevant medication | Continuosly from enrollment to 72h post.
  The continuous intake of the following drugs as chosen by discretion of the clinical staff is extracted from digital PDMS: Norepinephrine, Epinephrine, Dobutamin, inodilatators (Milrinon, Enoximon, Levosimendan)
Trop | at hours 0,6,12,24,48,72 post establishment of extracorporal membrane oxygenation (ECMO)
  The serum levels of troponine T will be compared between intervention and control group
CK | at hours 0,6,12,24,48,72 post establishment of extracorporal membrane oxygenation (ECMO)
  The Plasma levels of creatinkinase will be compared between intervention and control group.
Myoglobine | at hours 0,6,12,24,48,72 post establishment of extracorporal membrane oxygenation (ECMO)
  The Serum levels of myoglobine will be compared between intervention and control group.
Hemoglobine | at hours 0,6,12,24,48,72 post establishment of extracorporal membrane oxygenation (ECMO)
  The total blood concentration of hemoglobine will be compared between intervention and control group.
Haptoglobine | at hours 0,6,12,24,48,72 post establishment of extracorporal membrane oxygenation (ECMO)
  The serum levels of haptoglobine will be compared between intervention and control group.
paO2 | at hours 0,6,12,24,48,72 post establishment of extracorporal membrane oxygenation (ECMO)
  The arterial partial pressure of oxygen as measured by point-of-care blood gas analysis is going to be compared between intervention and control group
paCO2 | at hours 0,6,12,24,48,72 post establishment of extracorporal membrane oxygenation (ECMO)
  The arterial partial pressure of carbon dioxide as measured by point-of-care blood gas analysis is going to be compared between intervention and control group.
SaO2 | at hours 0,6,12,24,48,72 post establishment of extracorporal membrane oxygenation (ECMO)
  The saturation of hemoglobine with oxygen in an arterial blood sample as measured by point-of-care blood gas analysis is going to be compared between intervention and control group.
SvO2 | at hours 0,6,12,24,48,72 post establishment of extracorporal membrane oxygenation (ECMO)
  The saturation of hemoglobine with oxygen in a central venous blood sample as measured by point-of-care blood gas analysis is going to be compared between intervention and control group.
Horowitz index | at hours 0,6,12,24,48,72 post establishment of extracorporal membrane oxygenation (ECMO)
  The Horowitz index, calculated as paO2/FiO2 is going to be compared between intervention and control group.
pH | at hours 0,6,12,24,48,72 post establishment of extracorporal membrane oxygenation (ECMO)
  The pH of an arterial blood sample is going to be compared between intervention and control group.
HCO3 | at hours 0,6,12,24,48,72 post establishment of extracorporal membrane oxygenation (ECMO)
  The levels of bicarbonate of an arterial blood sample are going to be compared between intervention and control group.
BE | at hours 0,6,12,24,48,72 post establishment of extracorporal membrane oxygenation (ECMO)
  The base excess of an arterial blood sample is going to be compared between intervention and control group.
N | at hours 0,6,12,24,48,72 post establishment of extracorporal membrane oxygenation (ECMO)
  The blood levels of sodium are going to be compared between intervention and control group.
K | at hours 0,6,12,24,48,72 post establishment of extracorporal membrane oxygenation (ECMO)
  The blood levels of potassium are going to be compared between intervention and control group.
C | at hours 0,6,12,24,48,72 post establishment of extracorporal membrane oxygenation (ECMO)
  The blood levels of chloride are going to be compared between intervention and control group.
Lactate | at hours 0,6,12,24,48,72 post establishment of extracorporal membrane oxygenation (ECMO)
  The blood levels of lactate are going to be compared between intervention and control group.
Mode of Ventilation | at hours 0,6,12,24,48,72 post establishment of extracorporal membrane oxygenation (ECMO)
  The mode of mechanical ventilation is going to be compared between intervention and control group
FiO2 | at hours 0,6,12,24,48,72 post establishment of extracorporal membrane oxygenation (ECMO)
  The inspiratory oxygen fraction at mechanical ventilation is going to be compared between intervention and control group
Peak inspiratory pressure (pmax) | at hours 0,6,12,24,48,72 post establishment of extracorporal membrane oxygenation (ECMO)
  The peak inspiratory pressure at mechanical ventilation is going to be compared between intervention and control group
PEEP | at hours 0,6,12,24,48,72 post establishment of extracorporal membrane oxygenation (ECMO)
  The positive end exspiratory pressure at mechanical ventilation is going to be compared between intervention and control group
Ventilation frequency | at hours 0,6,12,24,48,72 post establishment of extracorporal membrane oxygenation (ECMO)
  The frequency of mechanical ventilation (cycles/min) is going to be compared between intervention and control group.
Tidal volume | at hours 0,6,12,24,48,72 post establishment of extracorporal membrane oxygenation (ECMO)
  The tidal volume achieved by mechanical ventilation is going to be compared between intervention and control group.
Total minute ventilation | at hours 0,6,12,24,48,72 post establishment of extracorporal membrane oxygenation (ECMO)
  The total minute ventilation as measured by the ventilation unit is going to be compared between intervention and control group.
Complicance | at hours 0,6,12,24,48,72 post establishment of extracorporal membrane oxygenation (ECMO)
  The airway compliance (c) as calculated from ventilator driving pressure(dp=pmax-PEEP) and tidal volume (V): c=V/dp is going to be compared between intervention and control group.
ASAT | at hours 0,6,12,24,48,72 post establishment of extracorporal membrane oxygenation (ECMO)
  The plasma levels of asparic acid aminotransferase will be compared between intervention and treatment group.
ALAT | at hours 0,6,12,24,48,72 post establishment of extracorporal membrane oxygenation (ECMO)
  The plasma levels of alanin aminotransferase will be compared between intervention and treatment group.
INR | at hours 0,6,12,24,48,72 post establishment of extracorporal membrane oxygenation (ECMO)
  The thrombin time as standardized international normal ratio will be compared between intervention and treatment group.
apTT | at hours 0,6,12,24,48,72 post establishment of extracorporal membrane oxygenation (ECMO)
  The activated partial thromboplastin time will be compared between intervention and treatment group.
Crea | at hours 0,6,12,24,48,72 post establishment of extracorporal membrane oxygenation (ECMO)
  The plasma creatinine concentration will be compared between intervention and treatment group.
eGFR | at hours 0,6,12,24,48,72 post establishment of extracorporal membrane oxygenation (ECMO)
  The glomerulary filtration rate, estimated from serum creatinine by the CKP-EPI formula will be compared between intervention and treatment group.
Volume status | at hours 0,6,12,24,48,72 post establishment of extracorporal membrane oxygenation (ECMO)
  For a clinical estimation of the renal function, the following parameters are extracted from the digital PDMS: Fluid intake, diuresis, additional loss of body fluids (e.g. gastral reflux, vomitting, extraction by kidney replacement therapy)
NSE | at hours 0,6,12,24,48,72 post establishment of extracorporal membrane oxygenation (ECMO)
  The serum levels of neuron specific enolase will be compared between intervention and treatment group.
Mortality | 30 days post enrollment
  Mortality within 30 days after enrollment due to any cause will be determined, if follow up is technically feasible

CONTACTS AND LOCATIONS:
Overall Officials: Jens Kubitz, Prof. Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Hospital Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adrie C, Laurent I, Monchi M, Cariou A, Dhainaou JF, Spaulding C. Postresuscitation disease after cardiac arrest: a sepsis-like syndrome? Curr Opin Crit Care. 2004 Jun;10(3):208-12. doi: 10.1097/01.ccx.0000126090.06275.fe. PMID 15166838
- [Background] Kellum JA, Song M, Venkataraman R. Hemoadsorption removes tumor necrosis factor, interleukin-6, and interleukin-10, reduces nuclear factor-kappaB DNA binding, and improves short-term survival in lethal endotoxemia. Crit Care Med. 2004 Mar;32(3):801-5. doi: 10.1097/01.ccm.0000114997.39857.69. PMID 15090965
- [Background] Peng ZY, Carter MJ, Kellum JA. Effects of hemoadsorption on cytokine removal and short-term survival in septic rats. Crit Care Med. 2008 May;36(5):1573-7. doi: 10.1097/CCM.0b013e318170b9a7. PMID 18434884
- [Background] Tomescu DR, Olimpia Dima S, Ungureanu D, Popescu M, Tulbure D, Popescu I. First report of cytokine removal using CytoSorb(R) in severe noninfectious inflammatory syndrome after liver transplantation. Int J Artif Organs. 2016 May 16;39(3):136-40. doi: 10.5301/ijao.5000489. Epub 2016 Apr 14. PMID 27079418
- [Background] Bruenger F, Kizner L, Weile J, Morshuis M, Gummert JF. First successful combination of ECMO with cytokine removal therapy in cardiogenic septic shock: a case report. Int J Artif Organs. 2015 Feb;38(2):113-6. doi: 10.5301/ijao.5000382. Epub 2015 Feb 3. PMID 25656010
- [Background] Bernardi MH, Rinoesl H, Dragosits K, Ristl R, Hoffelner F, Opfermann P, Lamm C, Preissing F, Wiedemann D, Hiesmayr MJ, Spittler A. Effect of hemoadsorption during cardiopulmonary bypass surgery - a blinded, randomized, controlled pilot study using a novel adsorbent. Crit Care. 2016 Apr 9;20:96. doi: 10.1186/s13054-016-1270-0. PMID 27059056

DOCUMENTS (1):
  • Study Protocol (2017-12-29): https://cdn.clinicaltrials.gov/large-docs/37/NCT03632837/Prot_000.pdf